CLINICAL TRIAL: NCT02952391
Title: Assessing Cholinergic Innervation in Parkinson's Disease Using the PET Imaging Marker [18F]Fluoroethoxybenzovesamicol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Teus van Laar, Prof. dr., University Medical Center Groningen
Other Study IDs: NL56173.042.15
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson's Disease
Keywords: cognition; cholinergic system
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Parkinson's disease patients: patients with Parkinson's disease, between the ages of 45 and 65, with a disease duration of 3 - 10 years
  Interventions: Other: [18F] FEOBV PET scan
- healthy control subjects: Healthy control subjects, between the ages of 45 and 65
  Interventions: Other: [18F] FEOBV PET scan

INTERVENTIONS:
Other: [18F] FEOBV PET scan — Cholinergic PET scan with the tracer [18F]Fluoroethoxybenzovesamicol

SUMMARY:
Although PD is considered predominantly as a motor disease caused by loss of dopaminergic neurons, multiple studies indicate that cholinergic dysfunction already starts in early PD and is crucial for the development of dementia in addition to motor symptoms.Because of its crucial role in CNS functioning and neurodegenerative disorders, including PD, it is of great importance to get a better understanding of the cholinergic functioning in the brain. Pathways of acetylcholine synthesis, transport and release provide possible targets for in vivo imaging of the cholinergic system. However,previous approaches are considered as indirect biomarkers of cholinergic terminal integrity because they measure both pre- and post-synaptic expressions. The novel vesicular acetylcholine transporter (VAChT) tracer [18F]Fluoroethoxy-Benzovesamicol ([18F]FEOBV) provides a more direct measurement of presynaptic cholinergic function. The use of [18F]FEOBV as a Positron Emission Tomography (PET) imaging marker of cholinergic innervations has, however, only been studied in healthy human volunteers and no data is available on patients.

With this study the differences in cholinergic function between PD patients and healthy aged-matched volunteers will be quantified. In addition the test-retest variability will be determined

DETAILED DESCRIPTION:
Rationale:

Cholinergic neurons play an important role in neurotransmission within the central nervous system (CNS). They are involved in complex functions like memory, learning, recognition, attention, consciousness, regulation of sleep-wake cycles and maintenance of posture and gait. Cholinergic neuron degeneration in the neocortex and hippocampus of the CNS, is an important neurochemical change observed in several neurodegenerative diseases, including Parkinson's disease (PD) and Alzheimer's disease (AD). Therefore, assessment of the vesicular acetylcholine transporter (VAChT) as an important molecular target in the cholinergic circuit, has sparked interest in the development of radiotracers for studying this target in vivo. Preclinical studies show the VAChT tracer (-)-5- [18F]Fluoroethoxybenzovesamicol ([18F]FEOBV) to be potentially useful in detecting cholinergic lesions in vivo. A previous [18F]FEOBV PET study confirms that the tracer binds to VAChT with the expected in vivo human brain distribution. The use of [18F]FEOBV as a PET imaging marker of cholinergic innervations has, however, only been studied in healthy human volunteers and no data is available on patients.

Objective:

The main objective of this study is to evaluate the differences in [18F]FEOBV binding between PD patients and healthy control subjects, in order to evaluate the clinical feasibility of [18F]FEOBV as a cholinergic imaging ligand in PD. Secondary objectives are the assessment of test-retest variability and confirming previous findings on [18F]FEOBV validation. Both secondary objectives are prerequisites for the main objective. In addition, an explorative analysis of the relationship between neuropsychological performance and cholinergic innervation will be performed.

Study design: In order to establish the difference in [18F]FEOBV binding between PD patients and healthy control subjects, the study will be conducted in three parts.

* The first part of the study is to establish [18F]FEOBV as a PET tracer for application in clinical research by confirming previous findings on [18F]FEOBV validation. This will include dynamic scanning of 3 healthy control subjects in 3 imaging sessions (0-120, 150-180, 210-240 min after injection of [18F]FEOBV). From this part of the study, the optimal short static scan period will be determined by comparing relative uptake values with the results of kinetic analysis.
* Part 2 of the study is to evaluate differences in [18F]FEOBV in Parkinson's disease and healthy controls. For this, the three dynamic scans of part 1 will be used and an additional 7 healthy control subjects and 10 PD patients will be included for a simple static scan (period determined after part 1 of the study).
* In part 3, test-retest variability is evaluated in both groups. Of each group, 5 patients will undergo a short second static scan.

All subjects will be screened within 30 days before the PET scan for demographic information and detailed clinical history.

Study population:

In total, 10 PD patients and 10 age matched control subjects will be included in the study, all between the ages of 45-65 years. Of the 10 control subjects, 3 will undergo full dynamic scanning, all other subjects included will undergo simple static scanning. A total of 10 subjects, 5 from each group, will undergo a second static scan. The patient group includes patients with Parkinson's disease with a disease duration of at least 3 years and maximum 10 years. All subjects will undergo a neuropsychological assessment.

Main study parameters/endpoints:

The main endpoint of this study is the difference in VAChT brain binding on a [18F]FEOBV PET-scan between PD patients and healthy control subjects.

Secondary endpoints are test-retest variability in both patients and healthy control subjects, and neuropsychological performance in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis Parkinson's disease (for patient group only)
* Disease duration between 3 and 10 years. (for patient group only)
* Age between 45 - 65 years
* Willingness to cooperate and sign written informed consent
* Able and fit enough to participate in this study

Exclusion Criteria:

* The refusal to be informed about an unforeseen clinical finding
* Pregnant women, breast feeding
* Participation in scientific research using radioactivity in the past 12 months , exceeding the maximum annual radiation dose
* Anticoagulant medication, antiplatelet agents used in the 5d before the imaging visit
* Contra-indication for MRI-scanning (metal parts in the body, red pigments in the skin as used in some tattoos)
* Other neurological conditions, more specifically neurodegenerative disorders and brain lesions.
* Treatment with deep brain stimulation
* prior history of neurologic or psychiatric illness (healthy control group only)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of subjects will be included in the study:
  * Patients with Parkinson's disease
  * Age-matched healthy control subjects A total of 20 subjects will be included in the study, with 10 subjects in each group.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
[18F]FEOBV binding | baseline
  the difference in VAChT brain binding on a [18F]FEOBV PET-scan between PD patients and healthy control subjects.

SECONDARY OUTCOMES:
Test-retest reliability | one week
  The percentage change in mean Standardized Uptake Value (SUV) between test and retest to assess test-retest variability.
Neuropsychological performance | baseline
  short neuropsychological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Teus van Laar, Prof. Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided